CLINICAL TRIAL: NCT00387868
Title: Phase II Study of Trimodality Therapy for Patients With Thymoma or Thymic Carcinoma at Significant Risk for Recurrence
Brief Title: Preoperative Treatment of Patients With High Risk Thymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHS07.0006a; NCT00509522 (obsolete NCT alias)
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Thymoma
Keywords: Thymoma; Thymic carcinoma; Preoperative chemotherapy and radiation; Response rate
MeSH Terms: conditions — Thymoma | interventions — Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Registration (Other): Cisplatin, Etoposide & concurrent radiotherapy
  Interventions: Drug: cisplatin and etoposide; Radiation: Concurrent Radiotherapy
- Surgical Resection (Other): No distant Progression post Registration Arm
  Interventions: Procedure: Surgical Resection
- Post Resection (Other): Assessment post surgical procedure to determine if at higher risk of recurrence or if complete resection could not be achieved.
  Interventions: Drug: cisplatin and etoposide

INTERVENTIONS:
Drug: cisplatin and etoposide — Cisplatin: 50mg/m2 - administered on days 1,8,29&36 Etoposide: 50 mg/m2 - administered on days 1-5 & 29-33
  Arms: Post Resection; Registration
Procedure: Surgical Resection — Resection will take place 4-8 weeks after completion of radiotherapy.
  Arms: Surgical Resection
Radiation: Concurrent Radiotherapy — Preoperative External Beam Radiotherapy
  Arms: Registration

SUMMARY:
This is a phase II study for patients with thymoma or thymic carcinoma thought to be at significant risk for recurrence following surgical removal. This study involves the use of combined chemotherapy and radiation therapy prior to surgery, in hopes of increasing the chances of complete resection. The chemoradiotherapy protocol is one which has been used extensively for other diseases, and the side effects are therefore well-documented. Patients with thymomas thought to be at significant risk for recurrence (by x-ray and pathology criteria) will be allowed to participate, and will undergo combined chemotherapy with radiation to the chest followed by surgical removal of the tumor and postoperative chemotherapy. The main outcome measured will be the rate of pathological complete response (e.g. no active tumor in the resected specimen) to the preoperative treatment. Patients will receive postoperative treatment based on surgical and pathologic criteria.

DETAILED DESCRIPTION:
Past experience has suggested that the ability to completely remove the thymoma using surgery is important in preventing recurrence. Strategies which would help the surgeon's ability to completely remove the tumor therefore need to be investigated.

This study represents a multi-institutional, phase II pilot trial of preoperative chemoradiotherapy followed by surgical resection and postoperative chemotherapy for patients with invasive thymoma or thymic carcinoma at significant risk for recurrence. We hypothesize that this strategy will be well-tolerated and produce response and resectability rates exceeding those previously published involving surgical resection alone, or preoperative chemotherapy followed by surgery. Patients with locally advanced thymoma, based on radiographic and biopsy criteria, will undergo pretreatment computed tomography (CT) scan and positron emission tomography (PET) followed by concurrent (simultaneous) chemotherapy (cisplatin and etoposide) and radiation. After this therapy, patients will be reassessed using computed tomography (CT) and PET, and undergo surgical resection of their tumors. Following resection, patients will be either observed, or treated with postoperative chemotherapy, or chemotherapy and radiation. Correlative genomic, serologic and pathologic studies will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven thymoma or thymic carcinoma.
* Invasive thymoma determined by specific radiographic criteria determined by CT scan.
* Acceptable kidney, liver, bone marrow, and respiratory functions.
* Karnofsy performance status greater than 80%.
* Patients must have a CT of the chest with IV contrast within 60 days of enrollment.
* Tumors larger than 8cm in greatest diameter on CT scan.
* For tumors 5-8cm in greatest diameter on CT scan, one or more of the following radiographic criteria must also be present on IV contrast CT Scan:
* Multifocal calcification
* Heterogeneous appearance
* Irregular of scalloped borders
* Obvious great vessel invasion or encirclement

Exclusion Criteria:

* Considered unable to medically tolerate surgical resection at the time of initial presentation.
* Radiographic evidence of stage IVA thymoma.
* Pretreatment biopsy showing WHO type A thymoma unless obvious great vessel invasion/encirclement is present on CT scan.
* Previous radiation therapy to the chest which would preclude the administration of radiation.
* Patents receiving other investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To determine the complete pathologic response rate to peroperative cisplatin and etoposide given concurrently with radiation in patients with thymoma thought to be at high risk for recurrence | 16 weeks

SECONDARY OUTCOMES:
Radiographic response to preoperative chemoradiotherapy by comparing pre and post treatment CT scans. | 16 weeks
Rate of complete resection following preoperative chemoradiotherapy as determined by pathologic examination of the specimen(s). | 1-5 weeks
Toxicities throughout the study treatment. | 5 years
The role of PET in predicting resectability, Masaoka stage and histologic type, as well as the response to preoperative chemoradiotherapy by comparing pre and post treatment PET scans | 10 years
Immunohistochemical assessment of relevant markers before and after chemoradiation (EGFR, p53,and Ki-67). | 10-12 years
Blood-based correlative studies: genetic polymorphisms (EGFR, DNA repair, inflammatory gene pathways) and serologic analysis (EGFR, VEGF, bFGF, pro-MMP2 levels) | 8-10 years
Recurrence rates and failure patterns following the treatment regimen. | 5-7 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Korst, MD, Principal Investigator — Valley Health Systems/ The Valley Hospital
Locations (2):
- Valley Health System - The Valley Hospital, Ridgewood, New Jersey, United States
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Korst RJ, Bezjak A, Blackmon S, Choi N, Fidias P, Liu G, Marx A, Wright C, Mock S, Rutledge JR, Keshavjee S. Neoadjuvant chemoradiotherapy for locally advanced thymic tumors: a phase II, multi-institutional clinical trial. J Thorac Cardiovasc Surg. 2014 Jan;147(1):36-44, 46.e1. doi: 10.1016/j.jtcvs.2013.08.061. Epub 2013 Oct 15. PMID 24139613
- [Derived] Wright CD, Choi NC, Wain JC, Mathisen DJ, Lynch TJ, Fidias P. Induction chemoradiotherapy followed by resection for locally advanced Masaoka stage III and IVA thymic tumors. Ann Thorac Surg. 2008 Feb;85(2):385-9. doi: 10.1016/j.athoracsur.2007.08.051. PMID 18222230